CLINICAL TRIAL: NCT02984618
Title: Gabriel Guimaraes: Sphenopalatine Block or Epidural Bloodpatch for Post Dural Puncture Headache: Randomized Controlled Trial
Brief Title: Sphenopalatine Block or Epidural Bloodpatch for Post Dural Puncture Headache: Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High recurrence of headache in SPG group.
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Substitute professor of Anesthesiology, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 60693416.0.0000.5558
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block; Blood Patch, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): Patients will receive sphenopalatine ganglion block with ropivacaine 0.375% 3ml on each side
  Interventions: Procedure: Sphenopalatine ganglion block
- Control group (Active Comparator): Patients will receive classic epidural blood patch with 20ml of autologous blood
  Interventions: Procedure: Epidural blood patch

INTERVENTIONS:
Procedure: Sphenopalatine ganglion block — Cotton- tipped applicators inserted up through the nose followed by infusion of ligdocaine through the applicators.
  Arms: Treatment group
Procedure: Epidural blood patch — Autologous sterile blood (20ml) will be infused in the lombar epidural space.
  Arms: Control group

SUMMARY:
Introduction: Recently sphenopalatine block emerged as an alternative to epidural blood patch for post dural puncture headache but the investigators do not know if it has significant efficacy when compared to epidural blood patch. Method: randomized trial where patients will randomly receive either sphenopalatine block or epidural blood patch. Pain relief to no pain or low intensity pain will be the main outcome

DETAILED DESCRIPTION:
Introduction: Recently sphenopalatine block emerged as an alternative to epidural blood patch for post dural puncture headache but the investigators do not know if it has significant efficacy when compared to epidural blood patch. Method: randomized clinical trial where patients with moderate to severe post dural puncture pain will randomly receive either sphenopalatine block or epidural blood patch. Pain relief to no pain or low intensity pain will be the main outcome. Pain recurrence, survival without pain and side effects (tinitus, low back pain, new dural puncture, sore throat) will be secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for post dural puncture headache
* Moderate to severe post dural puncture headache

Exclusion Criteria:

* Procedure failures: new dural puncture on epidural blood patch trial, unable to find epidural space, intolerance to insertion of nasal swabs.
* Follow up loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Pain relief | Pain reduction to no pain or low pain within 30 minutes of the intervention.
  Pain assessed by categorical verbal scale (no pain, low pain, moderate pain or severe pain) 30 minutes after the procedure.

SECONDARY OUTCOMES:
Tinitus | Incidence (dichotomic) of tinutus within 24 hours after the procedure.
Low back pain | Incidence (dichotomic) of low back pain within 24 hours after the procedure.
Sore throat | Incidence (dichotomic) of sore throat within 24 hours after the procedure.

OTHER OUTCOMES:
Pain relief survival | Incidence of new headache onset during the first two weeks
  Patients will be contacted for the first two weeks for monitoring new headache onsets.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimaraes, MsC, MD, Principal Investigator — Universidade de Brasilia
Locations (1):
- Hospital Universitário de Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No